CLINICAL TRIAL: NCT06056219
Title: Effects of Rhythmic-Based Training with Immersive Mirror Visual Feedback on Sensorimotor Function of Upper Extremity
Brief Title: Rhythmic-Based Training with Immersive Mirror Visual Feedback for Neuro-Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-ER-112-174
Record Dates: First submitted 2023-09-17; First posted 2023-09-28 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Rehabilitation; Virtual Reality; Mirror Movement Therapy
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirror therapy using a mirror box (Active Comparator): 30 minutes' exercise of mirror therapy followed by 20 minutes' task-oriented training
  Interventions: Device: Mirror therapy; Other: Task-oriented training
- Virtual reality-based mirror therapy with rhythmic skill training (Experimental): 30 minutes' activity of virtual reality-based mirror therapy with rhythmic skill training followed by 20 minutes' task-oriented training
  Interventions: Device: Virtual reality-based mirror therapy with rhythmic skill training; Other: Task-oriented training

INTERVENTIONS:
Device: Mirror therapy — 30 minutes' mirror therapy included movements of forearm, wrist, fingers and thumb, as well as a tendon gliding exercise of less-affected upper extremity using a mirror box
  Arms: Mirror therapy using a mirror box
Device: Virtual reality-based mirror therapy with rhythmic skill training — 30 minutes' virtual reality-based mirror therapy with rhythmic skill training included musical exercises involving virtual drums playing with less-affected upper extremity, and synchronized virtual drums playing and singing activity
  Arms: Virtual reality-based mirror therapy with rhythmic skill training
Other: Task-oriented training — 20 minutes' motor training targeted to goals that are relevant to the functional needs of the patient

SUMMARY:
In the proposed study, the investigators assumed that rhythmic-based training with immersive mirror visual feedback will provide a better treatment effects than traditional mirror therapy for the patients with unilateral stroke. The aim of the study is to examine the difference in the treatment effects among the combination of task-oriented training with either rhythmic-based training with immersive mirror visual feedback, or mirror therapy on the upper extremity function and brain activity of the stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke with unilateral side involved;
* A score of Mini-mental state examination greater than 24 for proving higher mental function
* Time of onset > 6 months before treatment begins; and
* Premorbid right-handedness.

Exclusion Criteria:

* Severe vision and hearing impairment;
* Major cognitive-perceptual deficit;
* Other brain disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Change in the result of Fugl-Meyer assessment (FMA) for motor function of upper extremity test | baseline, 9 weeks and 21 weeks
  Each item is rated on a three-point ordinal scale (2 points for the detail being performed completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The motor performance score ranges from 0 to 66 for the upper extremity.

SECONDARY OUTCOMES:
Change in the result of Box and block test | baseline, 9 weeks and 21 weeks
  The score is the number of blocks carried from one box to the other in one minute. Higher values represent a better outcome. The minimum and maximum value is 0 and 150 respectively.
Change in the result of Modified Ashworth scale (MAS) | baseline, 9 weeks and 21 weeks
  Muscle tone is defined by the resistance of a muscle being stretched without resistance. The MAS scores were distributed across the entire scale, ranging from 0 to 4, that is convenient for the clinician use. The grading of the scale is described as below: 0) no increase in muscle tone; 1) minimal resistance at the end of the range of motion (ROM); 1+) slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the reminder (less than half) of the ROM; 2) more marked increase in tone but only after part is easily flexed; 3) considerable increase in tone; and 4) passive movement is difficult and affected part is rigid in flexion or extension.
Change in the result of Semmes-Weinstein monofilament (SWM) test | baseline, 9 weeks and 21 weeks
  The Semmes-Weinstein monofilament test examines the cutaneous pressure threshold, range from 1.65-6.65. Higher values represent a worse outcome
Change in the result of Motor Activity Log | baseline, 9 weeks and 21 weeks
  Semi-structured interview examine how much and how well the subject uses their more-affected arm for 30 activities of daily living. Score range from 0-5. Higher values represent a better outcome

OTHER OUTCOMES:
functional Magnetic Resonance Imaging | baseline, 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No